CLINICAL TRIAL: NCT07125157
Title: Effect Of Task-Specific Training With And Without Biofeedback On Balance And Risk Of Falls In Chronic Ischemic Stroke Patients Of Central Lahore, Pakistan, A Randomized Controlled Trial
Brief Title: Effect Of Task-Specific Training With And Without Biofeedback On Balance And Risk Of Falls In Chronic Ischemic Stroke Patients Of Central Lahore, Pakistan
Acronym: TST-BIO-STROKE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Record submitted under wrong account; no participants enrolled
Sponsor: Syed Ali Behram Subazwari (Other)
Collaborators: Lincoln University College Malaysia (Other)
Responsible Party: Sponsor-Investigator, Syed Ali Behram Subazwari, Principal Investigator, Lincoln University College
Organization: Lincoln University College (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LUC/Ethc/Admin/SP/004/726
Record Dates: First submitted 2025-08-08; First posted 2025-08-15 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Chronic Ischemic Stroke; Balance Impairment; Risk of Fall
Keywords: stroke rehabilitation; biofeedback; task specific training; balance training; fall prevention; berg balance scale; time up and go
MeSH Terms: interventions — Biofeedback, Psychology

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two groups: one receiving task-specific training with biofeedback and the other receiving task-specific training without biofeedback.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be blinded to group allocation. Due to the nature of the intervention, therapists and participants cannot be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Task-Specific Training with Biofeedback (Experimental): Participants in this group will receive task-specific training combined with biofeedback. The intervention will focus on functional activities that challenge balance and mobility, while real-time feedback will be provided to improve motor control and postural stability. Training will be conducted under supervision for a set duration and frequency over the intervention period.
  Interventions: Behavioral: Task-Specific Training with Biofeedback
- Task-Specific Training without Biofeedback (Active Comparator): Participants in this group will receive the same task-specific training protocol without biofeedback. Functional tasks will be practiced to enhance balance and reduce fall risk. Training will be identical in duration and intensity to the experimental group but will not include feedback mechanisms.
  Interventions: Behavioral: Task-Specific Training without Biofeedback

INTERVENTIONS:
Behavioral: Task-Specific Training with Biofeedback — Participants in this group will undergo task-specific training focused on improving balance and reducing fall risk. Real-time biofeedback (e.g., visual or auditory cues) will be integrated into the training to enhance motor learning and postural adjustments. Sessions will be supervised and conducted multiple times per week over the intervention period.
  Other Names: Biofeedback-assisted task training
  Arms: Task-Specific Training with Biofeedback
Behavioral: Task-Specific Training without Biofeedback — Participants will receive task-specific training aimed at improving balance and fall prevention without any biofeedback assistance. The same set of functional exercises and session frequency will be followed as in the experimental group, ensuring the only difference is the absence of feedback stimuli.
  Other Names: Conventional task training
  Arms: Task-Specific Training without Biofeedback

SUMMARY:
This randomized controlled trial aims to evaluate the effects of task-specific training with and without biofeedback compared to conventional physical therapy on balance and fall risk in chronic ischemic stroke patients in Lahore, Pakistan. Sixty-six participants will be randomly allocated into three groups: Group 1 (task-specific training with biofeedback), Group 2 (task-specific training without biofeedback), and Group 3 (conventional physical therapy). The intervention will span 12 weeks, consisting of 36 sessions. Key outcome measures include the Berg Balance Scale, Timed Up and Go Test, and the Barthel Index. Assessments will be conducted at baseline, post-intervention, and three-month follow-up. The study hypothesizes that the use of biofeedback in task-specific training will produce significantly greater improvements in balance and reduced fall risk compared to conventional rehabilitation strategies. The study is being conducted at Shadman Medical Center in Lahore and is part of a PhD project from Lincoln University College.

DETAILED DESCRIPTION:
This randomized controlled trial investigates the comparative effectiveness of task-specific training with biofeedback, without biofeedback, and conventional physical therapy in improving balance and reducing fall risk among chronic ischemic stroke patients. The study consists of 66 participants, randomly assigned to three groups. Group 1 receives task-specific training using the Motor Relearning Program (MRP) principles, augmented with virtual reality-based biofeedback. Group 2 follows the same task-specific training without biofeedback. Group 3 receives conventional physical therapy following standard post-stroke rehabilitation protocols.

Participants will undergo 36 treatment sessions over a 12-week period, with three one-hour sessions per week. All interventions are delivered by qualified physiotherapists at the Department of Neurological and Functional Rehabilitation, Shadman Medical Center, Lahore.

Outcomes will be assessed using the Berg Balance Scale (BBS), Timed Up and Go (TUG) test, and the Barthel Index (BI) at baseline, post-intervention, and a 3-month follow-up. Randomization will be computer-generated, with blinding applied to assessors and data analysts.

The primary objective is to examine whether task-specific training with biofeedback significantly improves dynamic and static balance and reduces fall risk more effectively than the other two methods. Data will be analyzed using SPSS v21.0, applying repeated measures ANOVA and Cohen's d for effect size. A p-value ≤ 0.05 will be considered statistically significant.

The study has received ethical approval from Lincoln University College and is conducted under informed consent. Results will contribute to doctoral research and be submitted for peer-reviewed publication and presentation at scientific forums.

ELIGIBILITY:
Inclusion Criteria:

Chronic ischemic stroke patients (more than 3 months after stroke) Both Male and Female Patients Patients of 40 or above years of age Patients with Burnstorm stage 3 or above.) Patients with good cognitive function (score of 20 or more on MMSE) Patients who can ambulate 10 m (with or without the assistive device)

Exclusion Criteria:

Patients undergoing concurrent therapy or treatment that could influence the effectiveness of this study will be excluded from participation Patients presenting with contraindications to rehabilitation, such as severe uncontrolled hypertension, uncontrolled diabetes, or unstable angina, will be excluded from the study.

Individuals with prior neurological impairments apart from stroke.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Balance performance as measured by Berg Balance Scale (BBS) | Baseline (T0), Post-intervention (12 weeks, T2), and Follow-up (3 months post-intervention, TX)
  The BBS will assess balance performance across 14 items related to functional tasks such as sitting, standing, reaching, and turning. It is a widely validated tool in stroke rehabilitation.

SECONDARY OUTCOMES:
Risk of falls as measured by the Timed Up and Go (TUG) test | Baseline, Post-intervention (12 weeks), and Follow-up (3 months)
  The TUG test measures functional mobility and fall risk. The time (in seconds) to rise from a chair, walk 3 meters, turn, return, and sit is recorded. Lower times indicate better mobility and lower fall risk.

CONTACTS AND LOCATIONS:
Overall Officials: Syed Ali Behram Subazwari, Phd physiotherapy, Principal Investigator — Lincoln University College Malaysia
Locations (1):
- Shadman Medical Center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No